CLINICAL TRIAL: NCT00178698
Title: A Phase II Clinical Trial of Cisplatin + Gemcitabine HCl (GEM) + Low-Dose Metronomic Interferon-a (IFN-a) Combined With Fever-Range Whole-Body Thermal Therapy (FR-WB-TT) in Patients With Metastatic/or Locally Advanced Malignancies (Small-Cell Lung Cancer, Neuroendocrine Cancer, Gastric Cancer)
Brief Title: Hyperthermia/Thermal Therapy With Chemotherapy to Treat Inoperable or Metastatic Tumors
Acronym: FR-WB-TT/che
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C Bull, M.D., The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-04-259
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Neuroendocrine Cancer; Small Cell Lung Cancer; Non-Small Cell Lung Cancer; Gastric Cancer
Keywords: thermochemotherapy; fever range whole body; cisplatin; gemcitabine; daily low dose interferon alpha
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms | interventions — Cisplatin; Gemcitabine; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Thermochemotherapy
  Interventions: Other: thermochemotherapy; Drug: Cisplatin, Gemcitabine, Interferon-a

INTERVENTIONS:
Other: thermochemotherapy — cisplatin 60 mg/m2 i.v. over 4 hours on day 1 gemcitabine 600 mg/m2 i.v. over 60 minutes on day 3 interferon-alpha 1 million international units s.c. daily for protocol duration
  Other Names: fever-range systemic thermal therapy
Drug: Cisplatin, Gemcitabine, Interferon-a — cisplatin 60 mg/m2 i.v. over 4 hours gemcitabine 600 mg/m2 i.v. over 1 hour interferon-alpha 100,000 i.u. s.c.daily fever-range whole-body thermal therapy to 40 oC (104 oF) for 6 hours duration
Other: thermochemotherapy — After hydration and anti-emetics, cisplatin 60 mg/m2 i.v. is given over 4 hours on day 1. Also on day 1, begin daily low-dose interferon-alpha 1 million international units s.c. On day 3, 36 hours after cisplatin infusion, induce fever-range whole-body thermal therapy to 40 oC (104 oF) for a duration of 6 hrs. When the target temperature of 40 oC is reached, gemcitabine 600 mg/m2 is administered i.v. over 60 minutes, and the temperature is maintained at plateau for a total of 6 hours. The cycle is repeated at 21 to 28 day intervals.

SUMMARY:
Thermal therapy (hyperthermia, or heat) increases chemotherapy cancer cell kill. By itself, thermal therapy can also kill cancer cells. Whole body thermal therapy is a systemic treatment; whole-body fever-range thermal therapy can safely treat cancer cells wherever they are throughout the entire body. In this study, we are testing the combination of fever-range heat treatment and chemotherapy to test 1) The response of three types of cancer (small-cell lung, neuroendocrine cancer, lung cancer, and gastric cancer) to the thermo-chemotherapy improves cancer response compared to the effect of only chemotherapy drugs in current use; 2) whether the thermo-chemotherapy treatment helps the person's own body fight the cancer cells; and 3) whether this treatment is safe and comfortable for the patient. This study does not offer heat treatment alone. Any patient with inoperable or metastatic small cell lung cancer, neuroendocrine cancer (any organ), gastric cancer, or lung cancer, can be treated with the Phase II protocol therapy; however, the patient will need to undergo selected medical tests to make sure this treatment would be safe for them.

DETAILED DESCRIPTION:
The treatment cycle begins with 6 hours of intravenous (IV) hydration followed by an infusion of the anti-cancer drug, Cisplatin. In addition, at the beginning of this treatment, you will begin low-dose Interferon-alpha that will continue for the entire duration of your participation in this study. The low-dose Interferon-alpha interrupts the division of cancer cells, kills blood vessels feeding the cancer, and slows tumor growth, and as well boosts the body's immunity against the cancer.

Thirty-six hours after the cisplatin infusion, you will be treated with fever-range thermal therapy (whole-body hyperthermia). The fever-range whole-body thermal therapy enhances the effect of chemotherapy drugs against the cancer, and is thought to also boost your own immune response against the cancer. When the core body temperature reaches 104oF (40oC), a 30-minute (IV) infusion of another chemotherapy drug, gemcitabine (Gemzar) is given. Cisplatin, low-dose interferon-alpha and gemcitabine are the only chemotherapy drugs used in this treatment protocol. No other chemotherapy drugs are allowed to be given under this treatment plan.

The fever-range whole-body heat treatment is performed while you are lightly sedated. With this type of sedation, you are awake and can talk during the treatment but you are not uncomfortable. This type of sedation method is used to reduce any discomfort of the 6-hour heat treatment procedure yet allows you to talk to the nurses.

Your body temperature is raised to 104oF (40oC) over a period of 60-120 minutes. When your body first reaches the target 104oF, we administer the gemcitabine chemotherapy over 60 minutes and continue to maintain the 104oF body temperature for six hours. At the conclusion of the six hours of thermochemotherapy, you will be cooled off to your normal body temperature, which takes about 30-45 minutes. The entire treatment lasts approximately 8 hours. After the treatment is completed, we will observe you for 2 to 12 hours to make sure you have tolerated the treatment.

You will continue the low-dose Interferon-alpha injections once weekly. Additionally, you will be given 5-10 days of Leukine (sargramostim, GM-CSF) injections beginning 3-5 days after receiving chemotherapy to help support your immune system by helping your body create more white blood cells, which are important in helping your body fight infection.

After treatment, you will need a complete blood count with platelet and differential count each week. These lab studies can be done at your own doctor's office or hospital as long as you make sure that the results are faxed to us. They can also be done in our clinic. We will see you again in approximately three to four weeks and the treatment cycle will be repeated.

We always attempt to perform at least two thermo-chemotherapy cycles. After the second treatment, CT and/or MRI scans are repeated to see if your cancer is smaller. These scans, along with a physical examination and the lab studies, are used to determine if additional heat treatments will be performed. Additional treatments continue based on how well your response to the treatment. There is no limit to the number of heat treatments a patient may have.

ELIGIBILITY:
Inclusion Criteria:

- Any patient with inoperable or metastatic small-cell lung cancer, neuroendocrine cancer (any organ), gastric cancer, of lung cancer are eligible for protocol treatment.

However the patient:

* Must not have metastasis to the brain
* Must be able to achieve positive results on preliminary tests
* Must have a good ECOG performance status

Exclusion Criteria:

* Metastasis to the brain
* Poor results on preliminary physiological tests
* a Poor ECOG performance status score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2002-07; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Tumor Response by RECIST criteria (CR+PR) | 5 years
Response Duration | 5 years
Survival | 5 years

SECONDARY OUTCOMES:
Toxicity | 5 years
Quality of Life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Bull, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States